CLINICAL TRIAL: NCT00683423
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Crossover Trial to Evaluate the Efficacy and Safety of BMS-741672 in Patients With Diabetic Neuropathic Pain
Brief Title: BMS-741672 for Diabetic Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MB114-006
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: BMS-741672
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-741672 — Tablets, Oral, 100 mg, once daily, 3 weeks
  Arms: A
Drug: Placebo — Tablets, Oral, 0 mg, once daily, 3 weeks treatment period, 2 weeks washout, and 2 weeks follow-up
  Arms: B

SUMMARY:
The purpose of the study is to determine whether BMS-741672 improves neuropathic pain in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetics with painful, distal, symmetrical, sensory-motor neuropathy attributed to diabetes, of at least 12 months duration
* Screening HbA1c of ≥ 7% and ≤ 10%
* BMI ≤ 40 kg/m2

Exclusion Criteria:

* Patients with clinically significant, progressive, or potentially unstable disease of any body system including cardiovascular, gastrointestinal, central nervous system (CNS), psychiatric, endocrine (other than diabetes), tuberculosis or renal
* Women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Reduction in weekly average pain score for BMS drug vs. placebo, computed from diary scores | recorded during the last 7 days of treatment in each period

SECONDARY OUTCOMES:
Other glycemic, vascular, and mechanism-based biomarkers will be measured | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (8):
  - University Clinical Investigators, Inc., Tustin, California
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Comprehensive Neurosciences, Inc., St. Petersburg, Florida
  - The Pain & Rehabilitation Clinic Of Chicago, Chicago, Illinois
  - Advanced Biomedical Research Of America, Las Vegas, Nevada
  - Physicians East P.A., Greenville, North Carolina
  - Neurology Center Of Ohio, Toledo, Ohio
  - Research Institute Of Dallas, P.A., Dallas, Texas

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx